CLINICAL TRIAL: NCT06489587
Title: Creatine Supplementation At Simulated Altitude
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Responsible Party: Principal Investigator, Todd Hagobian, Chair and Professor, California Polytechnic State University-San Luis Obispo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-233
Record Dates: First submitted 2024-06-25; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-07

CONDITIONS: Exercise Performance
MeSH Terms: interventions — Creatine

STUDY DESIGN:
Intervention Model Description: Randomized study to two arms: 1) creatine supplementation, 2) glucose supplementation
Who Masked: Outcomes Assessor
Masking Description: Research staff collecting data will be masked to intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Supplementation (Active Comparator): Participants given Placebo (20 grams of glucose) daily in 5-gram servings (4 capsules), 4 times per day for 2 days.
  Interventions: Dietary Supplement: Placebo
- Creatine Supplementation (Experimental): Participants given Creatine (20 grams of glucose) daily in 5-gram servings (4 capsules), 4 times per day for 2 days.
  Interventions: Dietary Supplement: Creatine

INTERVENTIONS:
Dietary Supplement: Placebo — Participants given 40 grams of glucose in total to be taken over 2 days, in 5-gram servings (4 capsules), 4 times per day.
  Arms: Placebo Supplementation
Dietary Supplement: Creatine — Participants given 40 grams of creatine in total to be taken over 2 days, in 5-gram servings (4 capsules), 4 times per day.
  Arms: Creatine Supplementation

SUMMARY:
Creatine supplementation has been shown to increase exercise performance at sea level. The goal of this study is to determine the effects of creatine supplementation on exercise performance at simulated altitude.

DETAILED DESCRIPTION:
Military personnel often encounter harsh environments such as high altitudes and hypoxic conditions, leading to significant constraints on their exercise capacity and performance. At sea-level creatine supplementation increases exercise performance; however no experimental studies have examined the effect of creatine supplementation at simulated altitude. The overall objective of this study is to investigate the effects of creatine supplementation on exercise performance, via a repeated sprints test (Wingate Test) after a 2-day supplementation period, compared to a placebo group.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old
* BMI 18.5 to 40 kg/m2
* Habitually active (>150 minutes per week of moderate-vigorous physical activity)

Exclusion Criteria:

* Pregnant or trying to become pregnant
* Recent use of creatine supplementation
* Supplemental allergies

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Gender criteria are:
  * Cisgender man (non transgender)
  * Cisgender woman (non transgender)
  * Transgender man
  * Transgender woman
Enrollment: 60 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Peak power | Change from baseline to 3 days
  Peak power is measured in watts.

SECONDARY OUTCOMES:
Body Weight | Change from baseline to 3 days
  Body weight is measured in kilograms.
Relative peak power | Change from baseline to 3 days
  Relative peak power is measured in watts per kilogram.
Mean power | Change from baseline to 3 days
  Mean power is measured in watts.
Relative mean power | Change from baseline to 3 days
  Relative mean power is measured in watts per kilogram.
Fatigue index | Change from baseline to 3 days
  Fatigue index is measured in watts per second.

CONTACTS AND LOCATIONS:
Overall Officials: Todd Hagobian, PhD, Principal Investigator — California Polytechnic State University-San Luis Obispo
Locations (1):
- California Polytechnic State University, San Luis Obispo, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Data and documentation will be available under a data-sharing agreement. Information shared with outside collaborators will link data to two unique study identifiers (de-Identified) to maintain participant anonymity, and outside researchers and the community will not be allowed to have access to participant names and confidential information.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Seven years after the date of the last participant completing the study.
Access Criteria: Contact PI and a date-sharing agreement will be created that provides for (1) a commitment to use the data for research purposes only; (2) a commitment to securing the data using appropriate computer technology (password protected and encrypted); (3) a commitment to destroying or returning the data after analyses are completed and (4) a commitment not to attempt to identify participants individually.
URL: http://healthresearch.calpoly.edu/

DOCUMENTS (1):
  • Study Protocol (2024-01-26): https://cdn.clinicaltrials.gov/large-docs/87/NCT06489587/Prot_000.pdf